CLINICAL TRIAL: NCT03183739
Title: ASP8062 Phase 1 Study - A Placebo-controlled, Single and Multiple Ascending Oral Dose Study in Non-elderly Healthy Japanese Male and Female Subjects -
Brief Title: Study to Evaluate the Safety and Tolerability of ASP8062 in Healthy Japanese Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 8062-CL-0004
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
Keywords: ASP8062; Pharmacokinetics; Safety
MeSH Terms: interventions — ASP8062

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ASP8062 lower dose (Experimental): Subjects will receive a single dose of ASP8062 on Day 1, followed by 5 days of washout (Days 2-6) and once daily dosing for 14 consecutive days (Days 7-20) at the same dose level.
  Interventions: Drug: ASP8062
- ASP8062 middle dose (Experimental): Subjects will receive a single dose of ASP8062 on Day 1, followed by 5 days of washout (Days 2-6) and once daily dosing for 14 consecutive days (Days 7-20) at the same dose level.
  Interventions: Drug: ASP8062
- ASP8062 higher dose (Experimental): Subjects will receive a single dose of ASP8062 on Day 1, followed by 5 days of washout (Days 2-6) and once daily dosing for 14 consecutive days (Days 7-20) at the same dose level.
  Interventions: Drug: ASP8062
- Placebo (Placebo Comparator): Subjects will receive a single dose of Placebo on Day 1, followed by 5 days of washout (Days 2-6) and once daily dosing for 14 consecutive days (Days 7-20) at the same dose level.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8062 — ASP8062 will be administered orally.
  Arms: ASP8062 higher dose; ASP8062 lower dose; ASP8062 middle dose
Drug: Placebo — Placebo will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and evaluate pharmacokinetics of single and multiple ascending oral doses of ASP8062 in nonelderly Japanese male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight at screening: ≥ 50.0 kg and < 80.0 kg for male, ≥ 40.0 kg and < 70.0 kg for female.
* Body Mass Index (BMI) at screening: ≥ 17.6 kg/m^2 and < 26.4 kg/m^2 [BMI = Body weight (kg) ÷ {Body height (m)^2}].
* Female subjects must agree to consistently use 2 forms of highly effective birth control starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subjects must not donate ova starting at informed consent and throughout the clinical study period, and for 28 days after the final study drug administration.
* Male subjects and female spouse/partners who are of childbearing potential must be using condom and one of the highly effective birth control starting informed consent throughout the clinical study period and for 90 days after final study drug, if vasectomy is not performed for male subjects.
* Male subjects must not donate sperm starting at informed consent and throughout the clinical study period, and for 90 days after study drug administration.

Exclusion Criteria:

* Subjects who participated or are scheduled to participate in any clinical trials or post-marketing studies within 120 days before screening test or during the screening test to the hospital admission (Day -2).
* Subjects who received or is scheduled to receive any medications (including over-the-counter drugs) within seven days before the hospital admission.
* Any deviation from the normal range of blood pressure, pulse, body temperature, or routine 12-lead ECG at screening or on the day of hospital admission (Day -1).
* Subjects who meet any of the criterion for laboratory tests at screening or on the day of hospital admission (Day -2).
* Any deviation from the normal range of routine 12-lead ECG at screening.
* Subjects with a complication or history of drug allergies.
* Subjects who developed upper gastrointestinal symptoms (nausea, vomiting, stomachache, etc.) within seven days before the hospital admission.
* Subjects with a history of gastrointestinal resection except for appendicitis.
* Subjects with a complication or history of hepatic disease, cardiac disease, respiratory disease, gastrointestinal disease, renal disease, endocrine disease, cerebrovascular disease or malignant tumor.
* Subjects who received ASP8062 previously.
* Subject has a relevant history of suicide attempt or suicidal behavior.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of adverse events | Up to Day 38
  Adverse events (AEs) will be coded using Medical Dictionary for Regulatory Activities (MedDRA).
Safety assessed by vital signs: supine blood pressure | Up to Day 38
  To assess the vital sign as a criteria of safety and tolerability variables.
Safety assessed by vital signs: supine pulse rate | Up to Day 38
  To assess the vital sign as a criteria of safety and tolerability variables.
Safety assessed by vital signs: axillary body temperature | Up to Day 38
  To assess the vital sign as a criteria of safety and tolerability variables.
Orthostatic challenge tests | Up to Day 20
  To assess the orthostatic challenge tests as a criteria of safety and tolerability variables.
Safety assessed by laboratory tests: Hematology | Up to Day 38
  To assess hematology as a criteria of safety and tolerability variables.
Safety assessed by laboratory tests: Biochemistry | Up to Day 38
  To assess biochemistry as a criteria of safety and tolerability variables.
Safety assessed by laboratory tests: Urinalysis | Up to Day 38
  To assess urinalysis as a criteria of safety and tolerability variables.
Safety assessed by 12-lead electrocardiogram | Up to Day 21
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Columbia-Suicide Severity Rating Scale | Up to Day 20
  To assess the suicide risk
Safety assessed by body weight | Up to Day 38
  To assess the body weight as a criteria of safety and tolerability variables.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter for ASP8062: Maximum observed concentration (Cmax) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
PK parameter for ASP8062: Time to maximum concentration (Tmax) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
PK parameter for ASP8062: Terminal elimination half-life (t1/2) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
PK parameter for ASP8062: Apparent total systemic clearance after single or multiple extra-vascular dosing (CL/F) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
PK parameter for ASP8062: Area under the concentration-time curve (AUC) from the time of dosing to 24 h after dosing (AUC24) | Up to Day 6
  To assess the PK of ASP8062 in single dose part.
PK parameter for ASP8062: AUC from the time of dosing extrapolated to time infinity (AUCinf) | Up to Day 6
  To assess the PK of ASP8062 in single dose part.
PK parameter for ASP8062: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to Day 6
  To assess the PK of ASP8062 in single dose part.
PK parameter for ASP8062: Time point prior to the time point corresponding to the first measurable (non-zero) concentration (tlag) | Up to Day 6
  To assess the PK of ASP8062 in single dose part.
PK parameter for ASP8062: Apparent volume of distribution during the terminal elimination phase after single extra-vascular dosing (Vz/F) | Up to Day 6
  To assess the PK of ASP8062 in single dose part.
PK parameter for ASP8062: AUC from the time of dosing to the start of the next dosing interval (AUCtau) | From Day 7 to Day 38
  To assess the PK of ASP8062 in multiple dose part.
PK parameter for ASP8062: Concentration immediately prior to dosing at multiple dosing (Ctrough) | From Day 7 to Day 20
  To assess the PK of ASP8062 in multiple dose part.
PK parameter for ASP8062: Percentage of AUCinf that is estimated by extrapolation (AUCinf (%extrap)) | Up to Day 6
  To assess the PK of ASP8062 in single dose part
PK parameter for ASP8062: Terminal elimination rate constant (Lambda z) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
PK parameter for ASP8062: Time of the last measurable concentration (tlast) | Up to Day 38
  To assess the PK of ASP8062 in single dose part and multiple dose part.
Accumulation Ratio (Rac) of Cmax | From Day 7 to Day 38
  To assess the PK of ASP8062 in multiple dose part.
Rac of AUC | From Day 7 to Day 38
  To assess the PK of ASP8062 in multiple dose part.
Peak-Trough Ratio for last dosing in multiple dose part | Day 20 and Day 21
  To assess the PK of ASP8062 in multiple dose part.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Sumida City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.